CLINICAL TRIAL: NCT06133309
Title: Phenomenological Explorations of the Esketamine-Induced Transient Dissociative State
Acronym: EXPEDIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-CHITS-008; 2023-A01528-37 (Other: Id-RCB)
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Depressive Disorder
Keywords: Depressive disorder; Experiential Phenomenological Interview; Eskétamine; Transient dissociative state; Consciousness contents
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Depressive patients (Experimental): Patients suffering from depressive disorder and treated with Esketamine between 2 days and 3 months prior to the study.
  Interventions: Behavioral: Experiential Phenomenological Interview

INTERVENTIONS:
Behavioral: Experiential Phenomenological Interview — Consciousness fluidity of patients suffering from depressive disorder and treated with Esketamine will be evaluated thanks to Experiential Phenomenological Interview and EQFC "Trait" questionnaire

SUMMARY:
Ketamine is an anaesthetic used in low doses to treat depressive disorders. A related molecule, Esketamine, has recently been launched on the market for the treatment of resistant depression. One of the side effects of ketamine, like Esketamine, is induction of transient dissociative state. Dissociation has been described as disruption in continuity of conscious thought and emotion, cognitive processes disorganisation and an alteration in self-perception and environment perception. A study of healthy volunteers receiving ketamine showed that this state was manifested by altered sensory perceptions, with increased noise sensitivity, visual distortions and altered time perception. Few studies have looked at this phenomenon in the Esketamine context. However, it is a frequent side effect. With ketamine, it has been shown that anxiety associated with dissociative experience reduces the antidepressant effect. Benzodiazepines use for anxiolytic purposes is also thought to limit the antidepressant effect.

It is necessary to explore the Esketamine induced transient dissociative state in order to clarify this state and develop therapeutic strategies. The investigators have chosen a phenomenological approach, which is the only way to evaluate consciousness contents and structures, in order to explore this state using the experiential phenomenological interview.

DETAILED DESCRIPTION:
Patients will be identified when they come for an Esketamine session performed as part of routine practice in the Psychiatry Department of Hôpital Sainte Musse. The clinician, who is also the study investigator, will then select patients who meet the protocol's inclusion criteria and inform them of the research before administering the Esketamine. He will explain the study in detail and give them the information letter.

Patients will then be seen again in consultation outside the Esketamine sessions, as part of routine practice, within a minimum of 48 hours. During this consultation, the investigating physician will obtain their oral consent to their participation in the research, resulting in a research consultation lasting around 45 minutes and including :

* an audio recording of an Experiential Phenomenological Interview;
* completion of the EQFC "Trait" questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed in the Psychiatry Department of Hôpital Sainte Musse, with depressive state characterized by the DSM-V criteria and treated with Esketamine between 2 days and 3 months prior to the study;
* Patient over the age of 18;
* Patient presented transient dissociative state during Esketamine treatment;
* Patient able to express his/her consent prior to participation in the study;
* Patient who understands and speaks French.

Exclusion Criteria:

* Patient with major anxiety and panic attack during an Esketamine-induced dissociative state, regardless of Esketamine effect;
* Patient under judicial protection (guardianship, curatorship...) or safeguard of justice;
* Pregnant, parturient or breast-feeding women;
* Any other reason that, in the opinion of the investigator, would interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Consciousness fluidity evaluation by Experiential phenomenological interviews | 1 day
  Qualitative assessment by Experiential phenomenological interviews.

SECONDARY OUTCOMES:
Consciousness fluidity evaluation by EQFC "Trait" questionnaire | 1 day
  Qualitative assessment by EQFC "Trait" questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel DIAS ALVES, MD PhD, Study Director — Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmes EA, Brown RJ, Mansell W, Fearon RP, Hunter EC, Frasquilho F, Oakley DA. Are there two qualitatively distinct forms of dissociation? A review and some clinical implications. Clin Psychol Rev. 2005 Jan;25(1):1-23. doi: 10.1016/j.cpr.2004.08.006. PMID 15596078
- [Background] McIntyre RS, Rosenblat JD, Nemeroff CB, Sanacora G, Murrough JW, Berk M, Brietzke E, Dodd S, Gorwood P, Ho R, Iosifescu DV, Lopez Jaramillo C, Kasper S, Kratiuk K, Lee JG, Lee Y, Lui LMW, Mansur RB, Papakostas GI, Subramaniapillai M, Thase M, Vieta E, Young AH, Zarate CA Jr, Stahl S. Synthesizing the Evidence for Ketamine and Esketamine in Treatment-Resistant Depression: An International Expert Opinion on the Available Evidence and Implementation. Am J Psychiatry. 2021 May 1;178(5):383-399. doi: 10.1176/appi.ajp.2020.20081251. Epub 2021 Mar 17. PMID 33726522
- [Background] Aust S, Gartner M, Basso L, Otte C, Wingenfeld K, Chae WR, Heuser-Collier I, Regen F, Cosma NC, van Hall F, Grimm S, Bajbouj M. Anxiety during ketamine infusions is associated with negative treatment responses in major depressive disorder. Eur Neuropsychopharmacol. 2019 Apr;29(4):529-538. doi: 10.1016/j.euroneuro.2019.02.005. Epub 2019 Feb 13. PMID 30772118
- [Background] Pereira S, Brennan E, Patel A, Moran M, Wallier J, Liebowitz MR. Managing dissociative symptoms following the use of esketamine nasal spray: a case report. Int Clin Psychopharmacol. 2021 Jan;36(1):54-57. doi: 10.1097/YIC.0000000000000327. PMID 32804743
- See also: EQFC Questionnaire — https://hal.science/hal-02074893/document